CLINICAL TRIAL: NCT00886600
Title: A Double-blind, Randomized, Parallel-group, Placebo-controlled Pilot Study to Investigate the Magnitude and Duration of Response and the Safety of MK0954 (50 mg Given Once or Twice Daily, or 100 mg Given Once Daily) Compared to Placebo Using Ambulatory Blood Pressure Monitoring
Brief Title: A Study to Investigate the Magnitude and Duration of Response of MK0954 Compared to Placebo in Patients With Hypertension (0954-021)(COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0954-021; MK0954-021; 2009_581
Record Dates: First submitted 2009-04-22; First posted 2009-04-23 (Estimated); Results first posted 2009-07-14 (Estimated); Last update posted 2015-08-27 (Estimated); Status verified 2015-08

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Losartan; Hydrochlorothiazide

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- 1 (Placebo Comparator): Placebo
  Interventions: Drug: Comparator: placebo; Drug: hydrochlorothiazide (HCTZ)
- 2 (Experimental): losartan 50 mg q.d.
  Interventions: Drug: losartan potassium; Drug: hydrochlorothiazide (HCTZ)
- 3 (Experimental): losartan 100 mg q.d.
  Interventions: Drug: losartan potassium; Drug: hydrochlorothiazide (HCTZ)
- 4 (Experimental): losartan 50 mg b.i.d.
  Interventions: Drug: losartan potassium; Drug: hydrochlorothiazide (HCTZ)

INTERVENTIONS:
Drug: losartan potassium — losartan potassium (50 or 100 mg) administered orally once daily (q.d.)or twice daily (b.i.d) for four weeks
  Other Names: MK0954
  Arms: 2; 3; 4
Drug: Comparator: placebo — placebo capsules to losartan potassium (50 or 100 mg) administered orally once daily (q.d.)or twice daily (b.i.d) for four weeks
  Arms: 1
Drug: hydrochlorothiazide (HCTZ) — open-label hydrochlorothiazide (HCTZ) 12.5 mg (for patients with Sitting Diastolic Blood Pressure (SiDBP) ≥85 mm Hg after 4 weeks of losartan monotherapy (Combination Therapy Period)) orally once daily (q.d.) for 2 weeks
  Other Names: HCTZ

SUMMARY:
The purpose of this study was to evaluate the magnitude and durations of the antihypertensive effects of losartan using ambulatory blood pressure monitoring (ABPM), and to evaluate the safety of losartan 50 and 100 mg doses compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Non-black men and women with mild to moderate hypertension and within 30% of their ideal body weight
* Patient is in good general health
* Blood pressure at time of randomization is 95-115 mm Hg

Exclusion Criteria:

* Secondary Hypertension or history of malignant hypertension
* History of stroke
* History of myocardial infarction
* Atrial flutter or atrial fibrillation
* History of congestive Heart failure
* Patient taking major psychotropic agent or anti-depressant
* Patient regularly uses NSAIDS or high dose aspirin
* Known positive test for HIV/AIDS or Hepatitis B
* Patient is being treated for acute ulcer disease
* Prior exposure to losartan
* Actively treated diabetes mellitus
* History of chronic liver disease
* Actively treated diabetes mellitus
* Any known bleeding or platelet disorder
* Absence of one kidney
* Women of childbearing potential
* Alcoholism or drug addiction

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 1991-05; Primary Completion 1992-05 (Actual); Study Completion 1992-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Weber MA, Byyny RL, Pratt JH, Faison EP, Snavely DB, Goldberg AI, Nelson EB. Blood pressure effects of the angiotensin II receptor blocker, losartan. Arch Intern Med. 1995 Feb 27;155(4):405-11. PMID 7848024

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited at 9 sites in the United States. Prime Therapy Period: May, 1991 to March, 1992.
Pre-assignment Details: Patients could be randomized if sitting diastolic blood pressure (SiDBP) after 2 and 4 weeks of placebo washout was 95-115 mm Hg and the difference between measurements at the 2 visits was ≤7 mm Hg. At the end of placebo baseline the mean 24-hr DBP using ambulatory blood pressure monitoring (ABPM) had to be at least 85 mm Hg.
Groups:
- Placebo / HCTZ 12.5 mg: Double-blind Monotherapy: Losartan placebo orally once daily for 4 weeks
  Combination Therapy Period: Losartan placebo + open-label hydrochlorothiazide (HCTZ) 12.5 mg (for patients with SiDBP ≥85 mm Hg after 4 weeks of losartan monotherapy) orally once daily for 2 weeks
- Losartan 50 mg q.d. / HCTZ 12.5 mg: Double-blind Monotherapy: Losartan 50 mg orally once daily (q.d.) for 4 weeks
  Combination Therapy Period: Losartan 50 mg + open-label HCTZ 12.5 mg (for patients with SiDBP ≥85 mm Hg after 4 weeks of losartan monotherapy) orally once daily for 2 weeks
- Losartan 100 mg q.d. / HCTZ 12.5 mg: Double-blind Monotherapy: Losartan 100 mg orally once daily (q.d.) for 4 weeks
  Combination Therapy Period:Losartan 100 mg once daily + open-label HCTZ 12.5 mg (for patients with SiDBP ≥85 mm Hg after 4 weeks of losartan monotherapy).orally once daily for 2 weeks
- Losartan 50 mg b.i.d. / HCTZ 12.5 mg: Double-blind Monotherapy: Losartan 50 mg orally twice daily (b.i.d.) for 4 weeks
  Combination Therapy Period: Losartan 50 mg twice daily + open-label HCTZ 12.5 mg (for patients with SiDBP ≥85 mm Hg after 4 weeks of losartan monotherapy) orally once daily for 2 weeks
Period: Double-blind Monotherapy
Arm/Group | Placebo / HCTZ 12.5 mg | Losartan 50 mg q.d. / HCTZ 12.5 mg | Losartan 100 mg q.d. / HCTZ 12.5 mg | Losartan 50 mg b.i.d. / HCTZ 12.5 mg
Started | 32 | 29 | 30 | 31
Completed | 30 | 28 (1 pt discontinued after Wk 4 due to AE starting in placebo baseline and continuing into double-blind) | 29 | 29
Not Completed | 2 | 1 | 1 | 2
Not completed — Adverse Event | 1 | 1 | 1 | 1
Not completed — Protocol Violation | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0
Period: Combination Therapy Period
Arm/Group | Placebo / HCTZ 12.5 mg | Losartan 50 mg q.d. / HCTZ 12.5 mg | Losartan 100 mg q.d. / HCTZ 12.5 mg | Losartan 50 mg b.i.d. / HCTZ 12.5 mg
Started | 28 (Patients did not continue from monotherapy period : 2-(Sitting Diastolic Blood Pressure (SiDBP) <85)) | 21 (Patients did not continue from monotherapy period : 4-(SiDBP <85); 3-(SiDBP ≥85)) | 21 (Patients did not continue from monotherapy period : 7-(SiDBP <85); 1-(SiDBP ≥85)) | 23 (Patients did not continue from monotherapy period : 5-(SiDBP <85); 1-(SiDBP ≥85))
Completed | 28 | 21 | 19 | 23
Not Completed | 0 | 0 | 2 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo / HCTZ 12.5 mg: Losartan placebo orally once daily for 4 weeks followed by Losartan placebo + open-label hydrochlorothiazide (HCTZ) 12.5 mg (for patients with SiDBP ≥85 mm Hg) orally once daily for 2 weeks
- Losartan 50 mg q.d. / HCTZ 12.5 mg: Losartan 50 mg orally once daily for 4 weeks followed by Losartan 50 mg + open-label HCTZ 12.5 mg (for patients with SiDBP ≥85 mm Hg) orally once daily for 2 weeks
- Losartan 100 mg q.d. / HCTZ 12.5 mg: Losartan 100 mg orally once daily for 4 weeks followed by Losartan 100 mg once daily + open-label HCTZ 12.5 mg (for patients with SiDBP ≥85 mm Hg).orally once daily for 2 weeks
- Losartan 50 mg b.i.d. / HCTZ 12.5 mg: Losartan 50 mg orally twice daily for 4 weeks followed by Losartan 50 mg twice daily + open-label HCTZ 12.5 mg (for patients with SiDBP ≥85 mm Hg) orally once daily for 2 weeks
- Total: Total of all reporting groups
Arm/Group | Placebo / HCTZ 12.5 mg | Losartan 50 mg q.d. / HCTZ 12.5 mg | Losartan 100 mg q.d. / HCTZ 12.5 mg | Losartan 50 mg b.i.d. / HCTZ 12.5 mg | Total
Number analyzed (Participants) | 32 | 29 | 30 | 31 | 122
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.2 (12.0) | 56.8 (12.1) | 51.2 (9.6) | 54.1 (9.0) | 53.5 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 10 | 9 | 13 | 39
  Male | 25 | 19 | 21 | 18 | 83
Race/Ethnicity [Number; unit: participants]
  Caucasian | 30 | 29 | 30 | 30 | 119
  Oriental | 0 | 0 | 0 | 1 | 1
  Filipino | 1 | 0 | 0 | 0 | 1
  Indian | 1 | 0 | 0 | 0 | 1
Diastolic 24-hr mean ambulatory blood pressure monitoring (ABPM) [Mean (Standard Deviation); unit: mm Hg] | 94.8 (5.9) | 94.0 (6.9) | 93.8 (6.0) | 94.4 (6.9) | 94.2 (6.4)
Sitting Diastolic Blood Pressure (SiDBP) [Mean (Standard Deviation); unit: mm Hg] | 100.7 (4.0) | 100.0 (4.6) | 101.5 (5.1) | 101.2 (4.8) | 100.9 (4.6)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in 24-hour Diastolic Ambulatory Blood Pressure Monitoring (ABPM) at Week 4
Time Frame: 24 hour period at Baseline and Week 4
Population: The efficacy analysis followed a "per protocol" approach in that only patients who completed the study according to the protocol were included in the analysis.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Placebo / HCTZ 12.5 mg | Losartan 50 mg q.d. / HCTZ 12.5 mg | Losartan 100 mg q.d. / HCTZ 12.5 mg | Losartan 50 mg b.i.d. / HCTZ 12.5 mg
Number analyzed (Participants) | 26 | 28 | 28 | 30
mm Hg | -0.2 (4.8) | -5.2 (5.1) | -6.4 (5.5) | -8.5 (6.7)

2. Primary Outcome: Mean Change From Baseline in 24-hour Systolic Ambulatory Blood Pressure Monitoring (ABPM) at Week 4
Time Frame: 24-hour period at baseline and Week 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Placebo / HCTZ 12.5 mg | Losartan 50 mg q.d. / HCTZ 12.5 mg | Losartan 100 mg q.d. / HCTZ 12.5 mg | Losartan 50 mg b.i.d. / HCTZ 12.5 mg
Number analyzed (Participants) | 26 | 28 | 28 | 30
mm Hg | 0 (7.8) | -9.2 (9.9) | -9.9 (7.6) | -13.2 (10.6)

3. Secondary Outcome: Mean Change From Baseline in Sitting Diastolic Blood Pressure (siDBP) 24 Hours After Morning Dose at Week 4
Time Frame: Baseline and 24-hours after morning dose at Week 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Placebo / HCTZ 12.5 mg | Losartan 50 mg q.d. / HCTZ 12.5 mg | Losartan 100 mg q.d. / HCTZ 12.5 mg | Losartan 50 mg b.i.d. / HCTZ 12.5 mg
Number analyzed (Participants) | 30 | 29 | 28 | 30
mm Hg | -2.1 (6.9) | -6.7 (7.8) | -9.6 (6.5) | -8.8 (7.8)

4. Secondary Outcome: Mean Change From Baseline in Sitting Diastolic Blood Pressure (siDBP) After Adding HCTZ 24 Hours After Morning Dose at Week 6
Time Frame: Baseline and 24-hours after morning dose at Week 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Placebo / HCTZ 12.5 mg | Losartan 50 mg q.d. / HCTZ 12.5 mg | Losartan 100 mg q.d. / HCTZ 12.5 mg | Losartan 50 mg b.i.d. / HCTZ 12.5 mg
Number analyzed (Participants) | 26 | 21 | 16 | 20
mm Hg | -4.6 (6.1) | -9.9 (6.3) | -10.7 (4.9) | -10.1 (7.8)

5. Secondary Outcome: Mean Change From Week 4 in Sitting Diastolic Blood Pressure (siDBP) Adding HCTZ 24 Hours After Morning Dose at Week 6
Time Frame: Baseline and 24-hours after morning dose at Week 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Placebo / HCTZ 12.5 mg | Losartan 50 mg q.d. / HCTZ 12.5 mg | Losartan 100 mg q.d. / HCTZ 12.5 mg | Losartan 50 mg b.i.d. / HCTZ 12.5 mg
Number analyzed (Participants) | 26 | 21 | 16 | 20
mm Hg | -4.0 (6.4) | -5.1 (7.8) | -4.0 (6.1) | -4.0 (6.9)

LIMITATIONS AND CAVEATS:
Safety has been reported in the literature.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.